CLINICAL TRIAL: NCT01904266
Title: Combined General Anesthesia Plus Paravertebral Block Versus General Anesthesia Plus Opioid Analgesia for Breast Cancer Surgery: A Prospective Randomized Trial
Brief Title: Paravertebral Blocks for Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00028824
Record Dates: First submitted 2013-06-03; First posted 2013-07-22 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Pain, Postoperative; Nerve Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GA + sham block (Sham Comparator): Patients will receive general anesthetic plus a sham paravertebral block
  Interventions: Procedure: GA + sham block
- GA + paravertebral block (Experimental): Patients will receive general anesthetic plus a paravertebral block
  Interventions: Procedure: GA + paravertebral block

INTERVENTIONS:
Procedure: GA + paravertebral block — 20 cc ropivacaine 0.2% will be administered in an ultrasound-guided paravertebral block
  Arms: GA + paravertebral block
Procedure: GA + sham block — Injection of 1 cc saline subcutaneously
  Arms: GA + sham block

SUMMARY:
This research project intends to look at the effect that a certain type of freezing injection, called a paravertebral block, has on the pain after an operation for breast cancer, the amount of pain relief that is needed and the side effects from this pain relief. The hypothesis is that the paravertebral block, in combination with a general anesthetic will reduce both pain scores and the amount of strong pain killers (opioids) that is needed. This will reduce the side effects of the pain killers such as nausea and vomiting.

This will be assessed by comparing it a general anesthetic with pain killers given through the intravenous (IV) as is routine practice. Patients requiring breast cancer surgery, who agree to be involved in the trial, will be randomly allocated into two groups: both groups will receive a block, then a standardised and optimised general anesthetic. In one group however the block is simply a small injection under the skin (a sham block), whereas the other group will receive a proper paravertebral block prior to this. Both groups will receive opioids as necessary, depending on both their bodies reaction during the surgery and their pain scores when they wake up.

The paravertebral block is a very safe procedure with a very low side effect profile, and many studies have shown a benefit in breast cancer surgery. The investigators would like to assess this in our own practice. The block is normally inserted under some light sedation, with freezing into the skin initially. It is normally very well tolerated. The sham block will also be performed under light sedation and freezing into the skin. The patients will not be able to tell whether they are having the sham block or the paravertebral block, because both are very well tolerated. There are no potential complications from the sham block.

DETAILED DESCRIPTION:
Background Surgery for breast cancer can lead to a number of issues in the perioperative period. Both acute and chronic post-surgical pain are commonly encountered problems, with evidence that the degree of acute pain influences the likelihood of chronic pain. Post-operative nausea and vomiting (PONV) are also common, given the predominantly female surgical population and the requirement for opioid analgesia.

Paravertebral block (PVB) is an effective means of providing analgesia for mastectomy. A recent meta-analysis5 suggested that there is considerable evidence that paravertebral blocks with or without a general anesthetic (GA) provide superior post-operative analgesia to breast surgery operations done with a GA alone. There is also a reduced need for rescue analgesia and reduced opioid-related side effects. The results of this meta-analysis may be influenced by publication bias, and the results are difficult to interpret because the lack of standardisation of technique (single level injection, multi-level injection or continuous blockade via a catheter inserted into the paravertebral space) and the variety of the type and dosage of the local anesthetics used for the PVB. The meta-analysis does suggest that PVB is an effective technique for mastectomy with a minimal complication rate.

In our institution, the most common form of analgesia for mastectomy patients is systemic opioid analgesia. However, in the last two years, single level PVBs have been used with increasing frequency and reliable success. This is due in part to the use of ultrasound-guidance for placement of the PVB, which is a relatively simple technique with a well-defined end-point. The investigators have been using 0.2% ropivacaine, which was only mentioned in one study of the meta-analysis and was used with a multiple injection technique. The majority of studies used 0.5% bupivacaine, and most of these studies used PVB as the sole anesthetic technique. The next most common local anesthetic used was ropivacaine 0.5%, and this was more frequently used with multi-level injections. As the investigators use a single level injection in combination with a GA, these studies are not completely relevant to our current practice.

In this study, the investigators will compare PVB using Ropivacaine 0.2% combined with a GA, to GA alone with systemic analgesia.

Purpose The purpose of this study is to compare GA with systemic analgesia to GA with PVB. The parameters examined will be pain scores, perioperative opioid analgesia requirement, and PONV. Complications of PVB will also be examined.

Hypothesis GA plus PVB will reduce pain scores at rest and on movement, the need for rescue analgesia, and the incidence of PONV.

Study population:

Patients with Breast Cancer listed for surgery at the University Hospital of Alberta and the Cross Cancer Hospital. The study will commence following ethical approval.

Power calculations are required to determine recruitment numbers.

Methods:

The study population will be identified by the breast surgeons in their clinic, and potential recruits will be provided with information regarding the study protocol and techniques on that day. Patient consent will be obtained by the investigating team (study coordinator or anesthesiologist) on the day of surgery. Randomisation of participants will also occur at this time.

For those randomised to the PVB group, a block will be placed under sedation by one of the Acute Pain Service experienced in paravertebral blocks. The sham block group will receive some subcutaneous saline under ultrasound guidance, mild sedation and local anesthetic skin infiltration. All patients will receive a standard GA and post-operative protocol.

Patients who do not wish to enrol in the study will receive a general anesthetic plus appropriate analgesia according to the operating room anesthesiologist. No data will be recorded, apart from the fact that they declined to take part in the study.

Primary outcome measures:

1. Post-operative analgesia requirement

Secondary outcome measures:

1. Maximum pain score in the 24 hours following surgery
2. Incidence of PONV requiring additional treatment.
3. Maximum pain score in recovery at rest and on shoulder abduction
4. Incidence of perioperative complications
5. Intraoperative opioid requirement

Safety Concerns:

Paravertebral blocks have been used for many years. Major complications are rare. The investigators hypothesise that ultrasound should reduce these complications further as anatomical structures are directly visualized.

Major concerns:

1. Pleural puncture and pneumothorax
2. Paravertebral hematoma
3. Intrathecal local anesthetic injection
4. Local anesthetic toxicity
5. Paravertebral infection

Minor concerns:

1. Block failure
2. Epidural spread of local anaesthetic
3. Low blood pressure
4. Horner's Syndrome
5. Injection site hematoma

Study Protocol

1. Paravertebral block The patient will be reviewed by the study investigator then moved to the block area.

   Paravertebral block will be sited following intravenous access, commencement of IV crystalloid, and standard patient monitoring. A time out will confirm side of surgery which will be marked.

   Sedation and oxygen will be commenced prior to insertion of the block. The patient will be positioned in the seated position with the side of surgery clearly marked. The level between the transverse processes of T2 and T3 will be identified using ultrasound, then injection of 1% lidocaine to skin. Tissue movement and hydrolocation will confirm block needle position, with anterior movement of the pleura being the end point. Once this is reached, 20cc of ropivacaine 0.2% will be injected. The patients will progress to the standard anesthetic protocol.
2. Sham block The patient will be taken to the block area, where the IV and monitors will be connected as usual. Sedation and oxygen will be commenced. The sham block will occur as described for the true paravertebral block, including injection of lidocaine to anesthetize the skin, except that a small amount of normal saline (volume of which will be left to the anesthesiologist's discretion) will be injected subcutaneously instead of injection of ropivacaine next to the nerve.

   On the operating table, routine plus Bispectral (BIS) monitoring will be attached. If no midazolam has been administered, 0.03mg/kg will be given intravenously (IV). Fentanyl 1 microgram per kilogram IV will be given. Propofol will be titrated to allow insertion of a laryngeal mask airway (LMA), unless intubation is necessary. This will be at the discretion of the operating room anesthetist. Propofol via pump will be given at 200mcg/kg/min, aiming for a BIS score between 35 and 50. Phenylephrine or ephedrine can be titrated as necessary to maintain a mean arterial blood pressure above 60, or greater than 75% of the starting mean pressure. Spontaneous ventilation with pressure support will be used to maintain an end tidal carbon dioxide level of less than 50mmHg. Fentanyl (25mcg boluses) will be titrated to a respiratory rate of 8 - 15 breaths per minute. Ketorolac 15mg and Ondansetron 4mg IV will be given unless contra-indicated.
3. Post-operative Protocol

   All patients will receive standard post-operative orders:

   Patients will receive tramacet 3 tablets PO. Morphine 2mg IV will be given every 5 minutes as required for pain reported on the Numeric Rating Scale (NRS) of greater than 5. If intolerant of morphine, hydromorphone 0.4mg IV will be used. Further Ondansetron 4mg followed by 2 doses of Dimenhydrinate 25mg will be given for nausea and/or vomiting. Oxygen will be used to maintain saturations greater than 93%.

   Acetaminophen 975mg 6 hourly and Ibuprofen 400mg with meals three times daily will be given.

   Failure of this regime to control pain will trigger the addition of rescue analgesia.

   Rescue analgesia:

   Tramadol - 50 - 100mg po Q6h prn Oxycodone 5 - 10mg po Q3h prn Hydromorphone - 1mg sc Q2h PRN The patients will be assessed prior to PARR discharge regarding their pain scores at rest and on movement, and again on the morning following surgery.
4. Data Collection Data will be collected on a study sheet. Information will be kept confidential with no patient identifiers on the form, apart from a study number. This will reference a list kept securely by the investigators containing the patients' ULI numbers.

The pre- and intra-operative data recorded will be: demographic (age, weight, height), the surgical procedure, the amount of fentanyl, ephedrine and phenylephrine and propofol used.

The recovery data recorded will be: the amount of morphine or hydromorphone required, any anti-emetics given, the maximum pain score in recovery at rest and on shoulder abduction.

After discharge from recovery, the data recorded will be: anti-emetic use, rescue analgesia use, maximum pain score in the first 24 hours at rest and on movement.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Listed for Total Mastectomy +/- Axillary Node Dissection, or Partial Mastectomy

Exclusion Criteria:

* Patient refusal or inability to give informed consent
* Any contraindication for paravertebral blockade: coagulopathy, severe respiratory disease, local infection, untreated severe hypovolemia
* Allergy to propofol, severe egg allergy, or allergy to local anaesthetic agents
* Mastectomy plus flap reconstruction
* Bilateral procedures

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Post-operative analgesia consumption | 24 hours post-surgery
  Amount of morphine consumed in the 24 hours following surgery will be recorded

SECONDARY OUTCOMES:
Post-operative pain | 24 hours post-surgery
  Pain in the 24 hours following surgery will be assessed using a VAS scale
Nausea/vomiting | 24 hours post-surgery
  Incidence of nausea and vomiting in the 24 hours following surgery will be recorded on a 4-point scale
Pain upon movement | Within half an hour of return to recovery room
  Maximum pain score will be recorded in recovery at rest and on shoulder abduction
Intraoperative opioid requirement | During surgery
  Opioid consumption during surgery will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Vilholm OJ, Cold S, Rasmussen L, Sindrup SH. The postmastectomy pain syndrome: an epidemiological study on the prevalence of chronic pain after surgery for breast cancer. Br J Cancer. 2008 Aug 19;99(4):604-10. doi: 10.1038/sj.bjc.6604534. PMID 18682712
- [Background] Poleshuck EL, Katz J, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for chronic pain following breast cancer surgery: a prospective study. J Pain. 2006 Sep;7(9):626-34. doi: 10.1016/j.jpain.2006.02.007. PMID 16942948
- [Background] Gartner R, Kroman N, Callesen T, Kehlet H. Multimodal prevention of pain, nausea and vomiting after breast cancer surgery. Minerva Anestesiol. 2010 Oct;76(10):805-13. PMID 20935616
- [Background] Karmakar MK. Thoracic paravertebral block. Anesthesiology. 2001 Sep;95(3):771-80. doi: 10.1097/00000542-200109000-00033. No abstract available. PMID 11575553
- [Background] Schnabel A, Reichl SU, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of paravertebral blocks in breast surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2010 Dec;105(6):842-52. doi: 10.1093/bja/aeq265. Epub 2010 Oct 14. PMID 20947592
- [Background] Shkol'nik LD, Vasil'ev VIu, Soboleva LV. [Multi-injection thoracic paravertebral anesthesia during breast cancer operations]. Anesteziol Reanimatol. 2006 Jul-Aug;(4):80-5. Russian. PMID 17061598